CLINICAL TRIAL: NCT03462602
Title: Randomized Clinical Trial for Evaluation of the Use of Nasogastric Tube Decompression After Pancreatic Surgery
Brief Title: Nasogastric Tube in Pancreatic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Renyi Qin, Clinical professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TJDBPS04
Record Dates: First submitted 2018-02-26; First posted 2018-03-12 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Nasogastric Tube Decompression; Pancreatic Surgery

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NGT group (Experimental): NGT group
  Interventions: Procedure: NGT group
- non-NGT group (Experimental): non-NGT group
  Interventions: Procedure: non-NGT group

INTERVENTIONS:
Procedure: NGT group — After induction of anesthesia, a 14- or 16-Fr single-lumen NGT was placed in all patients. Its intragastric position was confirmed by intraoperative palpation. Randomization to the NGT or non-NGT group was performed on completion of surgery by computer-generated randomization provided by the supervision department.The NGT was retained until the return of bowel function (passage of flatus or passage of stool) in the patients assigned to the NGT group.
  Arms: NGT group
Procedure: non-NGT group — After induction of anesthesia, a 14- or 16-Fr single-lumen NGT was placed in all patients. Its intragastric position was confirmed by intraoperative palpation. Randomization to the NGT or non-NGT group was performed on completion of surgery by computer-generated randomization provided by the supervision department.The NGT was removed in the operation room immediately after the surgery in those assigned to the non-NGT group.
  Arms: non-NGT group

SUMMARY:
Introduction: The value of routine nasogastric tube (NGT) decompression after pancreatic surgeries is not yet established. Previous studies in the setting of abdominal surgery suggested that the use of NGT does not accomplish any of its intended goals.

Methods/design: This is a prospective, randomized, controlled multicenter trial with two treatment arms. One group underwent pancreatic surgeries with routine NGT and was left in place after surgery until the patient passed flatus or stool. The other group underwent pancreatic surgeries without receiving NGT decompression, in which the NGT was removed at the end of surgery.

Discussion: Routine NGT decompression after pancreatic surgeries does or does not appear to have its anticipated advantages would be discovered in this RCT.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age between 18 - 80 years.
* Patients underwent any kind of pancreatic surgeries, including but not limited to PD, distal pancreatectomy, central pancreatectomy, pancreatic enucleation, etc.
* Patients accepted the trial and could completed a written consent.

Exclusion Criteria:

* Combined with digestive tract obstruction before the surgery.
* History of upper abdominal surgery.
* Serious heart, brain, lung, metabolic diseases history.
* Pregnant women.
* Unwillingness or inability to consent for the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2020-05-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Time to flatus | 24 months
  It's described as the time patients to get flatus after operation

SECONDARY OUTCOMES:
Pulmonary complication | 24 months
  It was confirmed by clinical symptoms and CXR
Wound infection | 24 months
  Superficial or deep surgical-site infections are both considered and should be reported in medical records. Superficial infections are considered when skin or subcutaneous tissue is involved, whereas deep infection is considered when extending into the fascial layer.
Anastomotic leak | 24 months
  Including any type of Anastomotic leak, pancreatic fistula, bile leakage, etc.
Incisional hernia | 24 months
  Hernia or separation that occurred through a surgical incision in the abdominal wall deriving either from laparotomy or trocar incisions. All available data will be considered from medical records.
Length of Stay | 24 months
  Define as the day after surgery to dismiss.
Gastric upset | 24 months
  Any symptoms described by the subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Renyi Qin, pHD, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided